CLINICAL TRIAL: NCT00616902
Title: Clinical Study Protocol M10-221 The PRIMO II Study: Paricalcitol Injection Benefits in Renal Failure Induced Cardiac Morbidity in Subjects With Chronic Kidney Disease (CKD) Stage 5
Brief Title: The PRIMO II Study: Paricalcitol Injection Benefits in Renal Failure Induced Cardiac Morbidity in Subjects With Chronic Kidney Disease (CKD) Stage 5
Acronym: PRIMO II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was prematurely terminated due to low enrollment
Sponsor: Abbott (Industry)
Collaborators: Massachusetts General Hospital (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-221; 2007-005092-33 (EudraCT Number)
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Kidney Disease (CKD) Stage 5; Hypertrophy, Left Ventricular
Keywords: Zemplar, paricalcitol, PRIMO II
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertrophy, Left Ventricular | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol Injection 4 mcg/mL (Active Comparator): Paricalcitol Injection 4 mcg/mL given intravenously 3 times per week during dialysis
  Interventions: Drug: paricalcitol injection 4 mcg/mL
- Placebo Injection 4 mcg/mL (Placebo Comparator): Placebo Injection 4 mcg/mL given intravenously three times a week during dialysis
  Interventions: Drug: Placebo Injection 4 mcg/mL

INTERVENTIONS:
Drug: paricalcitol injection 4 mcg/mL — Paricalcitol Injection 4 mcg/mL intravenously three times a week during dialysis
  Other Names: ABT-358; paricalcitol; Zemplar
  Arms: Paricalcitol Injection 4 mcg/mL
Drug: Placebo Injection 4 mcg/mL — Placebo Injection 4 mcg/mL given intravenously three times a week during dialysis
  Other Names: placebo
  Arms: Placebo Injection 4 mcg/mL

SUMMARY:
To evaluate the effects of paricalcitol injection on cardiac structure and function over 48 weeks in subjects with Stage 5 Chronic Kidney Disease (CKD) receiving hemodialysis who have left ventricular hypertrophy (LVH).

ELIGIBILITY:
Inclusion Criteria:

* Stage 5 CKD receiving chronic hemodialysis three times per week for >= 3 months and <= 12 months from date of Randomization (Day 1).
* Serum intact parathyroid hormone (iPTH) value between 100-350 pg/mL.
* Serum calcium level between 8.4-10.5 mg/dL (2.1-2.6 mmol/L).
* Phosphate < 7 mg/dL.
* Serum albumin >= 3.0 g/dL (30 g/L).
* Echocardiogram results:

  * For females, left ventricular (LV) ejection fraction >= 50% and septal wall thickness between 11-17 mm.
  * For males, LV ejection fraction >= 50% and septal wall thickness between 12-18 mm.
* If the subject is receiving Renin Angiotensin-Aldosterone System (RAAS) inhibitors, the dose must have been stable for greater than one month prior to the Screening Period.
* A technically adequate baseline cardiac magnetic resonance imaging (MRI).
* If female, subject is not breast feeding or is not pregnant, or is not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile, or is of childbearing potential and practicing one of the following methods of birth control:
* Double-barrier method
* Hormonal contraceptives for at least three months prior to and during study drug administration
* Maintains a monogamous relationship with a vasectomized partner
* Total abstinence from sexual intercourse during the study.

Exclusion Criteria:

* Subject has previously been on active vitamin D therapy (calcitriol, paricalcitol, doxercalciferol, alfacalcidol) for a total duration greater than three months since the start of dialysis.
* Subject has a history of an allergic reaction or significant sensitivity to paricalcitol or to drugs similar to the study drug.
* Subject is expected to receive an increased dose of RAAS inhibitor (Angiotensin converting enzyme inhibitor [ACEi], Angiotensin II receptor blocker [ARB] or aldosterone inhibitor) during the course of the study.
* Subject has clinically significant coronary artery disease (CAD) within 3 months prior to the Screening Period, defined as one of the following:

  * Hospitalization for myocardial infarction (MI) or unstable angina; or
  * New onset angina with positive functional study or coronary angiogram revealing stenosis; or
  * Coronary revascularization procedure.
* Subject has major cardiac valve abnormality linked with left ventricular hypertrophy (LVH) and/or diastolic dysfunction, defined as one of the following:

  * Aortic valve area <= 1.5 cm2 or a mean gradient of > 20 mmHg; or
  * Regurgitation lesions; more than moderate mitral regurgitation or more than moderate aortic regurgitation.
* Subject has asymmetric septal hypertrophy.
* Subject has had a severe cerebrovascular accident (CVA) within the last three months (e.g., hemorrhagic) prior to screening.
* Full remission from a malignancy for less than one year except completely excised non-Melanoma skin cancer (e.g. basal or squamous carcinoma) or any history of bone metastasis.
* Subject has co-morbid conditions.
* Subject has received any investigational drug within 30 days prior to study drug administration or is currently enrolled in another clinical trial.
* Subject has poorly controlled hypertension.
* Subject has history of renal artery stenosis, primary aldosteronism or pheochromocytoma
* Subject is taking calcitonin, bisphosphonates, cinacalcet, glucocorticoids (except topical or inhaled glucocorticoids)
* Subject is currently receiving immunosuppressant therapy and/or high doses of glucocorticoids
* Subject is known to be HIV positive.
* Use of known inhibitors or inducers of cytochrome P450 3A (CYP3A) within two weeks prior to study drug administration
* Subject is contraindicated for the MRI examination
* Investigator considers subject unsuitable for any reason
* Subject has a history of drug or alcohol abuse within six months prior to screening
* Subject weighs more than 340 pounds (154 kg)
* Subject has had a liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Andress, MD, Study Director — Abbott
Locations (75):
- United States (29):
  - Arizona Kidney Disease & Hypertension Center, Phoenix, Arizona
  - Southwest Kidney Institute, Tempe, Arizona
  - National Institute of Clinical Research, Bakersfield, California
  - National Institute of Clinical Research, Los Angeles, California
  - University of Southern California Kidney Center, Los Angeles, California
  - North American Research Institute - California Kidney Specialist, San Dimas, California
  - Kidney Center of Simi Valley, Simi Valley, California
  - Western Nephrology and Metabolic bone disease, Arvada, Colorado
  - Western Nephrology, Westminster, Colorado
  - Washington Nephrology Associates, LLP, Washington D.C., District of Columbia
  - Fresenius Dialysis - Carrollwood, Tampa, Florida
  - FMC-NA Central Atlanta, Atlanta, Georgia
  - University of Illinois at Chicago - Nephrology Research, Chicago, Illinois
  - The University of Chicago - Stony Island Dialysis Unit, Chicago, Illinois
  - Evanston Northwestern Healthcare Corp. - Division of Nephrology, Evanston, Illinois
  - Research By Design, LLC, Evergreen Park, Illinois
  - North Suburban Nephrology, Gurnee, Illinois
  - Biolab Research LLC, Rockville, Maryland
  - Fresenius Medical Care, Kalamazoo, Michigan
  - V.A. Medical Center Research, Kansas City, Missouri
  - Washington University School of Medicine - Division of Renal Disease, St Louis, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - Brookdale Physicians Dialysis Associates, Brooklyn, New York
  - Nephrology Associates, PLLC, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - G. Edward Newman, MD, LLC, Knoxville, Tennessee
  - V.A. Tennessee Valley Healthcare System, Nashville, Tennessee
  - Southwest Houston Research, Ltd, Houston, Texas
  - The University of Texas - Health Science Center at San Antonio, San Antonio, Texas
- Australia (4):
  - Liverpool Hospital - Renal Unit, Liverpool, New South Wales
  - Westmead Hospital - Dept. of Renal Medicine, Sydney, New South Wales
  - The Princess Alexandra Hospital - Nephrology Dept., Wooloongabba, Queensland
  - Royal Melbourne Hospital - Dept. of Nephrology, Parkville, Victoria
- Czechia (5):
  - Faculty Hospital Brno, Brno
  - FN Pizen Lochotin - Charles University Teaching Hospital, Pizen
  - 1st LF UK - Nephrology Dept., Prague
  - IKEM - Nephrology Dept., Prague
  - 1st LF UK - Nephrology Dept. Strahov, Prague
- Germany (5):
  - KfH Nierenzentrum, Coburg
  - Gemeinschaftspraxis Dialyse, Dortmund
  - Gemeinschaftspraxix Karlstrasse, Düsseldorf
  - Niren-, Dochdruck und Dialysepraxis, Nettetal
  - Würzburg
- Greece (2):
  - IASO General - Renal Unit, Athens
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Italy (4):
  - Bologna
  - Monza
  - Pavia
  - Trieste
- Poland (4):
  - Katowice
  - Lodz
  - Szczecin
  - Warsaw
- Puerto Rico (2):
  - Fresenius Medical Care, Caguas
  - University of Puerto Rico, Rio Piedras
- Romania (5):
  - Spitalul "Dr. C. Davila" - Clinica de Nefrologie, Bucharest
  - Institut Clinic Fundeni - Clinica Medicine Interna/Nefrologie, Bucharest
  - Nefromed Dialysis Centre Cluj, Cluj-Napoca
  - Spitalul Clinic Judetean Cluj - Clinica de Nefrologie, Cluj-Napoca
  - Spitalul Clinic "Dr. C. I. Parhon" - Clinica de Nefrologie, Iași
- Russia (3):
  - City Clinical Hospital #52, Moscow
  - Moscow City Clinical Hospital named after Botkin, Moscow
  - Hospital for War Veterans #2, Moscow
- Spain (5):
  - Servicio de Nefrologia - Planta Baja, Córdoba
  - Fundacion Jimenez Diaz - Servicio de Nefrologia, Madrid
  - Hospital Universitario Son Dureta, Palma de Mallorca
  - Clinica Universitaria de la Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio - Servicio de Nefrologia, Seville
- Taiwan (4):
  - Cheng Hsin Rehabilitation Medical Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
  - Hsin-Jen Hospital, Xinzhuang
- United Kingdom (3):
  - University Hospitals Coventry and Warwickshire NHS Trust - University Hospital (UHCW), Coventry
  - Hammersmith Hospital, London
  - Salford Royal NHS Foundation Trust - Dept. of Nephrology, Salford

REFERENCES:
- [Derived] Thadhani R. Targeted ablation of the vitamin D 1alpha-hydroxylase gene: getting to the heart of the matter. Kidney Int. 2008 Jul;74(2):141-3. doi: 10.1038/ki.2008.219. PMID 18591942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 220 participants were to be randomized in a 1:1 ratio to each treatment group to receive paricalcitol injection or placebo at 75 US and ex-US sites. A stratified randomization scheme was used to ensure balance among treatment groups with respect to country, sex, and baseline Renin Angiotensin-Aldosterone System (RAAS) inhibitor use.
Pre-assignment Details: The Screening Period consisted of 3 visits and occurred within 6 weeks prior to participant randomization and enrollment into the Treatment Period of the study. For enrollment, all screening labs and echocardiogram requirements had to be met. Also, a technically adequate cardiac MRI had to be obtained for participant to be randomized into study.
Groups:
- Placebo Injection 4 Mcg/mL: Placebo Injection 4 mcg/mL given intravenously 3 times per week during dialysis.
Period: Overall Study
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Termination of study | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Number; unit: participants]
  < 40 years | 1 | 0 | 1
  40 - < 60 years | 3 | 2 | 5
  >= 60 years | 2 | 4 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 54.5 (16.01) | 58.8 (7.05) | 56.7 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in the Echocardiographic Assessment of Diastolic Function Assessed by Evaluating Changes in Diastolic Mitral Annular Relaxation Velocity (E') Over 48 Weeks.
Description: Mitral Annular relaxation velocity is a measure of diastolic heart function.
Time Frame: Baseline, 24 Weeks, and 48 Weeks/Early Termination
Population: The Intent-To-Treat (ITT) population - all randomized participants who were administered at least one dose of study drug. None of the participants completed 24 or 48 weeks.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline in Left Ventricular Mass Index (LVMI) Over 48 Weeks Measured by Cardiac Magnetic Resonance Imaging (MRI)
Description: Change from Baseline in left ventricular mass index (LVMI) over 48 weeks measured by cardiac MRI. The effects of paricalcitol injection on progression or regression of left ventricular hypertrophy (LVH) in participants with Stage 5 chronic kidney disease (CKD) on hemodialysis (HD) compared to placebo. Left Ventricular Mass is normalized to the participant's height by the following equation to obtain LVMI: LVM (g) divided by height (m)2.7.
  The primary comparison was between the 4 mcg paricalcitol injection and the placebo treatment groups in the change from baseline to Week 48.
Time Frame: Baseline, 24 Weeks, and 48 Weeks/Early Termination
Population: The Intent-To-Treat (ITT) population - all randomized participants who were administered at least one dose of study drug and the Evaluable population (a subset of ITT population and consists of those participants who have completed Week 24 visit). None of the participants completed 24 or 48 weeks.
Measure: Mean (Standard Deviation); unit: g/m2.7
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Evaluating Changes in the Additional Measure of Diastolic Function of Isovolumetric Relaxation Time (IVRT) Over 48 Weeks.
Description: Isovolumetric relaxation time is a measure of diastolic heart function.
Time Frame: Baseline, 24 Weeks, and 48 Weeks/Early Termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Evaluating Changes in the Additional Measure of Diastolic Function of Peak E-wave Velocity to Lateral E-wave Velocity (E/E') Over 48 Weeks.
Description: The ratio of peak E-wave velocity to lateral e-wave velocity is a measure of diastolic heart function.
Time Frame: Baseline, Week 24, and Week 48/Early Termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Evaluating Changes in the Additional Measure of Diastolic Function E-wave Deceleration Time (DT) Over 48 Weeks
Description: E-wave deceleration time is a measure of diastolic heart function.
Time Frame: Baseline, 24 Weeks, and 48 Weeks/Early Termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Biological Marker Triiodothyronine (T3).
Description: Plasma T3 is a circulating hormone that may have an effect on diastolic heart function and its level may be affected by treatment with paricalcitol. The study was terminated early (prior to any subject reaching Week 24). The values are for Baseline and Early Termination only. Each of the 12 randomized subjects terminated at different study weeks; therefore Early Termination cannot be defined as a specific week and varies for different subjects. Of the 12 subjects, 11 had early termination visits and 1 didn't. The final visit week range is 4-16.
Time Frame: Baseline and Early Termination Visit (4 Weeks, 5 Weeks, 7 Weeks, 8 Weeks, 14 Weeks, and 16 Weeks)
Population: The Intent-To-Treat (ITT) population - all randomized participants administered at least one dose of study drug. Results reported are from the early termination visit analysis for the subjects who terminated prematurely. None of the participants completed 24 or 48 weeks.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 5 | 6
nmol/L | 0.005 (0.5455) | -0.152 (0.3640)

7. Secondary Outcome: Change From Baseline in Biological Marker Plasma Troponin-T Over 48 Weeks
Description: Plasma troponin-t is a marker of heart damage and and its level may be affected by treatment with paricalcitol. The study was terminated early (prior to any subject reaching Week 24). The values are for Baseline and Early Termination only. Each of the 12 randomized subjects terminated at different study weeks; therefore Early Termination cannot be defined as a specific week and varies for different subjects. Of the 12 subjects, 11 had early termination visits and 1 didn't. The final visit week range is 4-16.
Time Frame: Baseline and Early Termination Visit (4 Weeks, 5 Weeks, 7 Weeks, 8 Weeks, 14 Weeks, and 16 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 5 | 6
mcg/L | -0.014 (0.0195) | -0.007 (0.0175)

8. Secondary Outcome: Change From Baseline in Biological Marker Plasma Interleukin-6 (IL-6) Over 48 Weeks
Description: Plasma IL-6 is a biomarker of inflammation that may have an effect on heart function and its level may be affected by treatment with paricalcitol. The study was terminated early (prior to any subject reaching Week 24). The values are for Baseline and Early Termination only. Each of the 12 randomized subjects terminated at different study weeks; therefore Early Termination cannot be defined as a specific week and varies for different subjects. Of the 12 subjects, 11 had early termination visits and 1 didn't. The final visit week range is 4-16.
Time Frame: Baseline and Early Termination Visit (4 Weeks, 5 Weeks, 7 Weeks, 8 Weeks, 14 Weeks, and 16 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 5 | 6
cm/sec | -0.200 (1.0954) | 0.333 (3.7771)

9. Secondary Outcome: Change From Baseline in Biological Marker Plasma High Sensitivity C-reactive Protein (hsCRP) Over 48 Weeks
Description: Plasma high sensitivity CRP is a biomarker of inflammation that may have an effect on heart function and its level may be affected by treatment with paricalcitol. The study was terminated early (prior to any subject reaching Week 24). The values are for Baseline and Early Termination only. Each of the 12 randomized subjects terminated at different study weeks; therefore Early Termination cannot be defined as a specific week and varies for different subjects. Of the 12 subjects, 11 had early termination visits and 1 didn't. The final visit week range is 4-16.
Time Frame: Baseline and Early Termination Visit (4 Weeks, 5 Weeks, 7 Weeks, 8 Weeks, 14 Weeks, and 16 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 5 | 6
mg/L | 1.104 (1.9361) | -0.762 (5.0013)

10. Secondary Outcome: Change From Baseline in Biological Marker Plasma B-Type Natriuretic Peptide (BNP)
Description: Plasma BNP is a product from the heart that becomes elevated with an enlarged heart and its level may be affected by treatment with paricalcitol. The study was terminated early (prior to any subject reaching Week 24). The values are for Baseline and Early Termination only. Each of the 12 randomized subjects terminated at different study weeks; therefore Early Termination cannot be defined as a specific week and varies for different subjects. Of the 12 subjects, 11 had early termination visits and 1 didn't. The final visit week range is 4-16.
Time Frame: Baseline and Early Termination Visit (4 Weeks, 5 Weeks, 7 Weeks, 8 Weeks, 14 Weeks, and 16 Weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Number analyzed (Participants) | 5 | 6
ng/L | -134.200 (119.6963) | 572.800 (903.6101)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Paricalcitol Injection 4 Mcg/mL | Placebo Injection 4 Mcg/mL
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol Injection 4 Mcg/mL (N=6) | Placebo Injection 4 Mcg/mL (N=6)
Chills (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was prematurely terminated due to low enrollment. Only 12 subjects were randomized at 10 investigative sites with none of the subjects completing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.